CLINICAL TRIAL: NCT01071603
Title: A Natural History Study of Tuberculosis in China; Correlates of a Successful Response to Treatment
Brief Title: Tuberculosis in China
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999910060; 10-I-N060
Record Dates: First submitted 2010-02-18; First posted 2010-02-19 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-01-29

CONDITIONS: Tuberculosis; Tuberculosis, Multidrug-Resistant; Extensively Drug Resistant Tuberculosis
Keywords: Biomarkers; Extrapulmonary TB; NTM; HRCT; MDRTB; Tuberculosis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Multidrug-Resistant; Extensively Drug-Resistant Tuberculosis; Tuberculosis, Extrapulmonary

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- In spite of well-researched treatments and therapies, 5 to 10 percent of tuberculosis (TB) patients who have initially successful TB treatments will relapse, usually within a year after completion of therapy. This percentage is even greater for patients who are infected with multi-drug resistant and extensively drug resistant types of TB. Because the People s Republic of China has the second highest number of TB cases in the world, researchers are interested in studying TB patients in China to evaluate their response to treatment on a long-term basis.

Objectives:

* To improve TB diagnosis and testing by determining the number and proportion of patients admitted with suspected TB who actually have TB (definite or probable).
* To assess the prevalence of non-tuberculosis bacteria among patients with presumed TB.

Eligibility:

- Individuals between 18 and 65 years of age who have been admitted to Henan Provincial Chest Hospital with suspected tuberculosis.

Design:

* Participants will be divided into three groups, based on their diagnosis after admission. Another group of individuals who do not have TB will be enrolled as controls for comparison purposes during the study.
* The study will use computed tomography (CT) scans of the chest at initial enrollment, 2 months, and 6 months to evaluate disease response to treatment. Incidents of TB that are not in the chest area (extrapulmonary TB) will also be studied.
* The study will also monitor the treatments and therapies used against the disease, changes in patients immune systems, and any changes in the biological samples taken over the course of treatment.

DETAILED DESCRIPTION:
Despite optimal antimicrobial treatment with directly observed short-course therapy (DOTS), about 5-10 percent of drug-compliant patients with cured tuberculosis (TB or MTB) relapse, usually within a year after completion of therapy. This percentage is even greater for patients that have previously been treated for TB who often are infected with multi-drug resistant (MDR) and extensively drug resistant (XDR) organisms. The People s Republic of China has the second highest number of cases of TB in the world, with a rate of 101 cases/100,000 person-years estimated for 2004. Based on the data of the 4th national TB epidemiological survey in 2000, it is estimated that there were 1.96 million instances of pulmonary TB. With an established MDR TB prevalence of 10.7 percent, there were an estimated 209,720 cases of pulmonary, bacteriology confirmed MDR TB in China in 2000. About half of all prevalent cases of TB disease in 2000 were extrapulmonary.

This prospective longitudinal natural history study will monitor 150 subjects with suspected TB at the Henan Provincial Chest Hospital during their initial response to antituberculous chemotherapy. The subjects will be divided into 3 groups of TB-infected individuals: Cohort A) acid-fast bacilli (AFB) smear positive pulmonary disease; Cohort B) smear negative pulmonary disease; and Cohort C) extra-pulmonary disease (EPTB) in order to reflect the spectrum of TB manifestations observed at Henan Provincial Chest Hospital. We will also be enrolling 45 non-TB suspects as controls (Cohort D). The control group will serve as a comparison group for exploratory immunologic and diagnostic assays that may, in the future, serve as ways to diagnose TB and/or evaluate response to therapy.

In this exploratory study, we will be looking at the change in total volume of disease as detected by computerized tomography scans of the chest at baseline, at 2 months, and at 6 months. We will also be looking at scanned regions of extrapulmonary TB. In addition, we will monitor chemotherapeutic regimen, changes in the host immune response, overall changes in clinical parameters, initial and acquired drug-resistance of the infecting isolates, and changes in bacterial and host markers in subject samples during chemotherapy. In each case, we will look for associations of these parameters with rates of disease resolution correlated with specific structural features determined by computerized tomography scanning of the sites of TB disease (with the exception of TB meningitis and cutaneous TB, for which there are no specific lesions to follow radiographically). These studies will allow us to evaluate the use of entry criteria in future clinical trials and eventual TB diagnosis confirmation using these entry categorizations. We will also be able to examine the impact of initial regimen selection, and subsequent modifications, mycobacterial strain characteristics, extent of disease, types of lesions and host immunologic response to the overall outcome of chemotherapy, as well as potentially identify surrogate markers for improving monitoring of the response to chemotherapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject must fulfill all inclusion criteria within his or her assigned cohort in order to be eligible to participate in this study.

Smear Positive TB (Cohort A)

* Age 18-65 years old
* Sputum AFB-smear positive (at least 1 positive smears out of 3) and exhibiting the signs or symptoms suggestive of pulmonary MTB disease
* If presently on anti-TB chemotherapy, having a regimen which started not more than 14 days prior to enrollment (please see note below)
* If previously treated for TB, having been off of anti-TB chemotherapy for at least 60 days before starting present regimen, or before enrollment if not presently on drugs
* Willingness to adhere to study visits and testing
* Willingness to have samples stored

Smear Negative TB (Cohort B)

* Age 18-65 years old
* Sputum AFB-smear negative (zero out of 3) and exhibiting the signs or symptoms suggestive of pulmonary MTB disease
* If presently on anti-TB chemotherapy, having a regimen which started not more than 14 days prior to enrollment (please see note below)
* If previously treated for TB, having been off of anti-TB chemotherapy for at least 60 days before starting present regimen, or before enrollment if not presently on drugs
* Willingness to adhere to study visits and testing
* Willingness to have samples stored
* Subjects with the above criteria who cannot expectorate and cannot produce sputum by induction

Extra Pulmonary TB (Cohort C)

* Age 18-65 years old
* Exhibiting the signs and symptoms suggestive of MTB EP disease

If presently on anti-TB chemotherapy, having a regimen which started not more than 14 days prior to enrollment (please see note below)

* If previously treated for TB, having been off of anti-TB chemotherapy for at least 60 days before starting present regimen, or before enrollment if not presently on drugs
* Willingness to adhere to study visits and testing
* Willingness to have samples stored

Controls (Cohort D):

* Age 18-65 years old
* No signs or symptoms of an active TB infection
* Willingness to adhere to study visit and testing
* Willingness to have samples stored

EXCLUSION CRITERIA:

A subject will be excluded from this study if he or she meets any of the following exclusion criteria from their assigned cohort. Also, potential participants may be excluded from the study on the basis of the investigator s judgment concerning the ability to comply with study procedures or posing an undue risk to the subject.

Cohort C Only

Evidence of pulmonary TB (If subject at enrollment is suspected to have both pulmonary TB and extrapulmonary TB, then s/he will be enrolled into Cohort A or B)

Cohort D (Controls)

* Those with signs or symptoms consistent with TB disease
* Women who report themselves to be pregnant or those found to be pregnant by a urine beta-HCG test during the protocol introduction and consent process;
* Those having a chest X-ray suggestive of active tuberculosis
* Use of immunosuppressive agents such as corticosteroids, TNF blocking agents, cyclosporine, methotrexate, or mycophenolate at entry
* Body mass index (BMI) <16
* History of systemic lupus erythematosus, rheumatoid arthritis, or other connective tissue disease
* The use of any of the following drugs within 30 days prior to study or anticipated use of these drugs within the next 60 days:
* Systemic cancer chemotherapy
* Systemic corticosteroids
* Immune globulin
* Interleukins
* Interferons
* Those with malignancies

Cohort A-C Scan Exclusions

The following will still be included in the study; however they will be excluded from the CT scanning (enrollment and follow-up) only:

* Those who are pregnant
* Those with a creatinine greater than 150 UL within 14 days of a scheduled CT scan (enrollment or follow-up)

Note that if subjects excluded by these above criteria for a study-related CT scan still require a CT scan because of medical necessity, the results of the CT scan will be collected by the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2010-02-02; Study Completion 2018-01-29

CONTACTS AND LOCATIONS:
Overall Officials: Clifton E Barry, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Henan Provincial Chest Hospital, Zhengzhou, China

REFERENCES:
- [Background] He GX, Zhao YL, Jiang GL, Liu YH, Xia H, Wang SF, Wang LX, Borgdorff MW, van der Werf MJ, van den Hof S. Prevalence of tuberculosis drug resistance in 10 provinces of China. BMC Infect Dis. 2008 Dec 11;8:166. doi: 10.1186/1471-2334-8-166. PMID 19077223
- [Background] Xianyi C, Fengzeng Z, Hongjin D, Liya W, Lixia W, Xin D, Chin DP. The DOTS strategy in China: results and lessons after 10 years. Bull World Health Organ. 2002;80(6):430-6. PMID 12131998
- [Background] Wallis RS. Surrogate markers to assess new therapies for drug-resistant tuberculosis. Expert Rev Anti Infect Ther. 2007 Apr;5(2):163-8. doi: 10.1586/14787210.5.2.163. No abstract available. PMID 17402829
- [Derived] Trauner A, Liu Q, Via LE, Liu X, Ruan X, Liang L, Shi H, Chen Y, Wang Z, Liang R, Zhang W, Wei W, Gao J, Sun G, Brites D, England K, Zhang G, Gagneux S, Barry CE 3rd, Gao Q. The within-host population dynamics of Mycobacterium tuberculosis vary with treatment efficacy. Genome Biol. 2017 Apr 19;18(1):71. doi: 10.1186/s13059-017-1196-0. PMID 28424085